CLINICAL TRIAL: NCT06777381
Title: Comparison of Post-Operative Pain Occurrence After Single Visit Root Canal Treatment with Two NiTi Rotary Files - a Randomized Clinical Trial
Brief Title: Comparison of Post-Operative Pain Occurrence After Single Visit Root Canal Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Amira lbrahim Mohamed, Researcher, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03460224
Record Dates: First submitted 2024-12-29; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: post-operative pain; ProTaper; M-Pro; single visit
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: ProTaper Universal system (Experimental): root canal treatment will be performed in single visit using ProTaper Universal system
  Interventions: Procedure: single visit root canal treatment using ProTaper Universal rotary system
- Group B: M-Pro rotary system (Experimental): root canal treatment will be performed in single visit using M-Pro rotary system
  Interventions: Procedure: single visit root canal treatment using M-Pro rotary system

INTERVENTIONS:
Procedure: single visit root canal treatment using ProTaper Universal rotary system — single visit endodontic treatment will be performed using ProTaper Universal rotary system for root canal preparation.
  Arms: Group A: ProTaper Universal system
Procedure: single visit root canal treatment using M-Pro rotary system — single visit endodontic treatment will be performed using MPro rotary systems for root canal preparation.
  Arms: Group B: M-Pro rotary system

SUMMARY:
The goal of this clinical trial is to compare the post-operative pain occurrence after single visit root canal treatment using Two NiTi Rotary Files. The main question it aims to answer is:

• Does an instrument design and instrumentation technique could affect postoperative pain incidence and intensity? Researchers will use ProTaper Universal rotary system or M-Pro rotary system for root canal preparation and compared postoperative pain intensity.

Participants will receive single visit endodontic treatment using either ProTaper or MPro systems for root canal preparation.

Participants will record Pain intensity at 24 hours and 7 days post-operative. Analgesics will be prescribed for the patients in need.

DETAILED DESCRIPTION:
The main cause of patient fear is expecting pain during root canal treatment. It is considered a major concern for dentists as well. During root canal preparation, periapical extrusion of pulpal tissue remnants, microorganisms or dentin chips may be one of the causes of postoperative pain. Depending on the fact that, instrument design and instrumentation techniques have an impact on the amount of extruded debris apically, many studies proved the ability of some rotary systems to reduce debris extrusion, permitting to achieve less pain sensation.

Therefore, the present clinical study aims to compare the postoperative pain intensity in molars with symptomatic irreversible pulpitis after single endodontic treatment visit using a full-sequence rotary Ni-Ti system either ProTaper or MPro systems Eighty patients with symptomatic irreversible pulpitis in mandibular first molars will be assigned into two groups. In group A (n=40): root canal preparation will be performed in single visit using ProTaper Universal system and in group B (n=40): root canal preparation will be performed in single visit using M-Pro rotary system. Pain intensity will be recorded by the patient using Numerical Rating Scale (NRS) at 24 hours and 7 days postoperative. Analgesics will be prescribed for the patients in case of need.

ELIGIBILITY:
Inclusion Criteria:

* Patient's diagnosis is symptomatic irreversible pulpitis in mandibular first molar.
* Males and females patients in a good health.
* Aged from 25 to 45 years old.
* Pulp vitality is confirmed with cold pulp test and an electric pulp test.

Exclusion Criteria:

* Pregnant females.
* Patients complaining from pain in more than one molar on the same side.
* Patients whose teeth react positively to percussion test.
* Patients who receive analgesics 12 hours before the start of the root canal treatment.
* Teeth having grade 2 or 3 mobility.
* Presence of periapical radiolucency or teeth with extra oral or intraoral sinus tract or fistula.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Record the intensity of postoperative pain after root canal treatment with ProTaper Universal and M-Pro endodontic rotary files. | 7 days
  Pain intensity will be recorded by the patient 24 hours and 7 days postoperatively. Pain assessment is evaluated using 10-point Numerical Rating Scale, where the endpoints are the extremes of no pain and worst pain. The severity of pain is assigned as follows: (0) equivalent to none/ (1) equivalent to slight pain / (2) equivalent to moderate pain and (3) equivalent to severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Clinic at Medical Research Centre of Excellence, National Research Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Khallaf ME, Aly Y, Mohamed AI. Comparison of post-operative pain prevalence after single visit endodontic treatment with two NiTi rotary files - a randomized clinical trial. Sci Rep. 2025 Dec 18;15(1):44128. doi: 10.1038/s41598-025-29029-8. PMID 41413418